CLINICAL TRIAL: NCT01266356
Title: A TMU/NIH Integrated Research Project Translation of Basic Research to Clinical Diagnosis and Treatment of Mild Traumatic Brain Injury (mTBI)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wen-Ta Chiu, Graduate Institute of Injury Prevention and Control, Taipei Medical University
Other Study IDs: 99019
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Traumatic Brain Injury
Keywords: Minor Traumatic Brain Injury; Translation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
This integrated research project is cooperated by an fully-experienced team of Taipei Medical University and National Institutes of Health. We hope that we can find out the disease of balance, anxiety and sick headaches through the translation of basic research to clinical diagnosis and treatment of Mild Traumatic Brain Injury (mTBI).

ELIGIBILITY:
Inclusion Criteria:

* willing to accept this research
* age above 17 years old
* brain injury patients who are in Glasgow Coma Scale(GCS) between 13 to 15

Exclusion Criteria:

* age under 16 years old
* serious brain injury patients
* pregnant women
* people who have accepted ears surgery once
* uremia
* Liver Cirrhosis

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Brain Injury Patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-08; Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ta Chiu, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan